CLINICAL TRIAL: NCT01154855
Title: Circulatory Microbial Components and Immune Regulators of Patients With Periodontal Disease and Rheumatoid Arthritis
Brief Title: Periodontal Disease and Circulatory Microbial Components
Acronym: CirCo
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, William Giannobile, Principal Investigator, University of Michigan
Other Study IDs: HUM00029568
Record Dates: First submitted 2010-03-16; First posted 2010-07-01 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Periodontal Disease
Keywords: Periodontal disease; Gum disease; Dental; Inflammation; Microorganisms; Bacteria
MeSH Terms: conditions — Periodontal Diseases; Gingival Diseases; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Dental plaque samples evaluated for microbial DNA
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Periodontitis: Patients with severe periodontal disease Intervention (Procedure/surgery): Prophylaxis; Gross debridement for diseased patients
  Other Names:
  Teeth cleaning
  1 per patient at 2nd visit lasting approximately 1 hour.
  Interventions: Procedure: Prophylaxis ; Gross debridement for diseased patients
- Healthy patients: Patients without periodontal (gum) disease Intervention (Procedure/surgery): Prophylaxis; Gross debridement for diseased patients
  Other Names:
  Teeth cleaning
  Interventions: Procedure: Prophylaxis ; Gross debridement for diseased patients

INTERVENTIONS:
Procedure: Prophylaxis ; Gross debridement for diseased patients — 1 per patient at 2nd visit lasting approximately 1 hour.
  Other Names: Teeth cleaning

SUMMARY:
The goal of this project is to study the immune activity of certain proteins present in the blood of patients with severe periodontal disease. Periodontal disease (gum disease) is the major cause of tooth loss among adults. Moderate to severe periodontal disease is reported to affect 5-15% of American adults. It begins with an infection of the tissues surrounding the teeth, and leads to a worsening inflammatory response. This study will aid in clarifying the way in which gum disease might affect certain systemic diseases.

DETAILED DESCRIPTION:
This project will have two specific goals: 1. Identify microorganism components in the serum of patients with severe periodontitis; and 2. Characterize the immune regulator activity of periodontitis serum. This proposed feasibility study will then aid in providing the support for an increased sample size and other design requirements for larger, more expanded human clinical trial testing.In this study, forty (40) subjects will be divided into 2 groups: 1) Healthy oral status group and 2) Severe periodontal disease. Patients will be clinically screened using standard periodontal measurements.

ELIGIBILITY:
Inclusion Criteria:

* 35 years or older
* Healthy patients or patients with severe periodontal disease
* Patients with or without Rheumatoid Arthritis
* Patients with at least 20 permanent teeth

Exclusion Criteria:

* Patients undergoing long-term (over 2 weeks) antibiotic-related therapy 3 months prior to study inclusion
* Patients receiving periodontal treatment 12 months prior to study inclusion (INCLUDING CLEANINGS)
* Patients will be excluded if they receive long-term use of medications known to affect periodontal status such as anti-inflammatory drugs, aspirin and ibuprofen
* Patients on immunosuppressive therapies, including glucocorticoids or cyclosporines, are excluded from participation in this study (inhalers are allowed)
* History of metabolic bone diseases such as rheumatoid arthritis or post-menopausal osteoporosis
* Pregnant women or women attempting to become pregnant

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 40 adult subjects comprised of two populations: 1) healthy (n=20) and 2) severe periodontal disease (n=20)
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Identify microorganism components in the serum of patients with severe periodontitis | 1hour
  microorganism components will be analyzed in serum samples collected before teeth cleaning and again 5 minutes after teeth cleaning

SECONDARY OUTCOMES:
Characterize the immune regulator activity of periodontitis serum | 1 hour
  microorganism components will be analyzed in serum samples collected before teeth cleaning and again 5 minutes after teeth cleaning

CONTACTS AND LOCATIONS:
Overall Officials: William V Giannobile, DDS, DMedSc, Principal Investigator — University of Michigan

REFERENCES:
- [Background] Akira S, Uematsu S, Takeuchi O. Pathogen recognition and innate immunity. Cell. 2006 Feb 24;124(4):783-801. doi: 10.1016/j.cell.2006.02.015. PMID 16497588
- [Background] Forner L, Nielsen CH, Bendtzen K, Larsen T, Holmstrup P. Increased plasma levels of IL-6 in bacteremic periodontis patients after scaling. J Clin Periodontol. 2006 Oct;33(10):724-9. doi: 10.1111/j.1600-051X.2006.00964.x. Epub 2006 Aug 10. PMID 16901299
- [Background] D'Aiuto F, Parkar M, Andreou G, Suvan J, Brett PM, Ready D, Tonetti MS. Periodontitis and systemic inflammation: control of the local infection is associated with a reduction in serum inflammatory markers. J Dent Res. 2004 Feb;83(2):156-60. doi: 10.1177/154405910408300214. PMID 14742655
- [Background] Garlet GP, Martins W Jr, Ferreira BR, Milanezi CM, Silva JS. Patterns of chemokines and chemokine receptors expression in different forms of human periodontal disease. J Periodontal Res. 2003 Apr;38(2):210-7. doi: 10.1034/j.1600-0765.2003.02012.x. PMID 12608917
- [Background] Pussinen PJ, Paju S, Mantyla P, Sorsa T. Serum microbial- and host-derived markers of periodontal diseases: a review. Curr Med Chem. 2007;14(22):2402-12. doi: 10.2174/092986707781745604. PMID 17896988
- [Result] Marchesan J, Jiao Y, Schaff RA, Hao J, Morelli T, Kinney JS, Gerow E, Sheridan R, Rodrigues V, Paster BJ, Inohara N, Giannobile WV. TLR4, NOD1 and NOD2 mediate immune recognition of putative newly identified periodontal pathogens. Mol Oral Microbiol. 2016 Jun;31(3):243-258. doi: 10.1111/omi.12116. Epub 2015 Sep 10. PMID 26177212